CLINICAL TRIAL: NCT06719570
Title: An Open-Label Study to Evaluate the Effect of a High-Fat Meal on the Pharmacokinetics of Doravirine/Islatravir (100 mg/0.25 mg) Fixed-dose Combination Tablet and to Compare the Pharmacokinetics of Doravirine/Islatravir to Doravirine and Islatravir Single Entities in Healthy Adult Participants
Brief Title: A Study of Doravirine and Islatravir as a Single Entity or Combination Therapy and the Effect of Food in Healthy Adult Participants (MK-8591A-055)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 8591A-055; MK-8591A-055 (Other: MSD); CA42943 (Other: Celerion)
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — doravirine; islatravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- MK-8591A Sequence 1A (Experimental): Participants will receive Doravine/Islatravir (DOR/ISL) fixed-dose combination (FDC) tablet under fasting conditions followed by a DOR/ISL FDC tablet under fed conditions followed by a single dose Doravine tablet and a single dose Islatravir capsule under fasting conditions.
  Interventions: Drug: MK-8591A; Drug: Islatravir; Drug: Doravine
- MK-8591A Sequence 2A (Experimental): Participants will receive DOR/ISL FDC tablet under fasting conditions followed by a single dose DOR tablet and a single dose ISL capsule under fasting conditions followed by DOR/ISL FDC tablet under fed conditions.
  Interventions: Drug: MK-8591A; Drug: Islatravir; Drug: Doravine
- MK-8591A Sequence 1B (Experimental): Participants will receive DOR/ISL FDC tablet under fed conditions followed by a DOR/ISL FDC tablet under fasting conditions followed by a single dose DOR tablet and a single dose ISL capsule under fasting conditions.
  Interventions: Drug: MK-8591A; Drug: Islatravir; Drug: Doravine
- MK-8591A Sequence 2B (Experimental): Participants will receive DOR/ISL FDC tablet under fed conditions followed by a single dose DOR tablet and a single dose ISL capsule under fasting condition followed by a DOR/ISL FDC tablet under fasting conditions.
  Interventions: Drug: MK-8591A; Drug: Islatravir; Drug: Doravine
- MK-8591A Sequence 1C (Experimental): Participants will receive a single dose DOR tablet and a single dose ISL capsule under fasting conditions followed by DOR/ISL FDC tablet under fasting conditions followed by followed by a DOR/ISL FDC tablet under fed conditions.
  Interventions: Drug: MK-8591A; Drug: Islatravir; Drug: Doravine
- MK-8591A Sequence 2C (Experimental): Participants will receive a single dose DOR tablet and a single dose ISL capsule under fasting conditions followed by DOR/ISL FDC tablet under fed conditions followed by followed by a DOR/ISL FDC tablet under fasting conditions.
  Interventions: Drug: MK-8591A; Drug: Islatravir; Drug: Doravine

INTERVENTIONS:
Drug: MK-8591A — Fixed dose combination tablet
  Other Names: Doravirine/Islatravir (DOR/ISL) Fixed-Dose Combination (FDC)
Drug: Islatravir — Oral capsule
  Other Names: MK-8591; ISL
Drug: Doravine — Oral tablet
  Other Names: MK-1439; DOR

SUMMARY:
The purpose of this study is to learn what happens to MK-8591A in a person's body over time. Researchers will compare what happens to MK-8591A in the body when it is given with and without food.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria include, but are not limited to:

* Has a body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m^2
* Is medically healthy with no clinically significant medical history, physical examination, clinical laboratory profiles, vital signs, and electrocardiograms (ECGs)

Exclusion Criteria:

Exclusion Criteria include, but are not limited to:

* Has a history or presence of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has a history of cancer (malignancy)

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Area under the curve from time 0-infinity (AUC0-inf) of DOR | At designated time points up to ~30 days
  AUC0-inf is a measure of plasma drug concentration from time 0 to infinity and is estimated as the area under the plot of plasma concentration against time 0 to infinity after drug administration. Blood samples collected at designated time points will be used to determine the AUC0-inf of DOR.
Area under the curve from time 0 to last measurable concentration (AUC0-last) of Doravine | At designated time points up to ~30 days
  AUC0-last is defined as the area under the concentration-time curve from time 0 to time of last measurable concentration of DOR. Blood will be collected at designated time points to determine the AUC0-last of DOR.
Maximum plasma concentration (Cmax) of doravine | At designated time points up to ~30 days
  Cmax is the maximum concentration of the drug observed in plasma. Blood samples collected at designated time points will be used to determine Cmax of DOR.
Plasma concentration at 24 hours postdose (C24) of DOR | At designated time points up to ~24 hours postdose
  C24 is the concentration at 24 hours postdose of the drug observed in plasma. Blood samples collected at 24 postdose will be used to determine C24 of DOR.
AUC0-inf of ISL | At designated time points up to ~30 days
  AUC0-inf is a measure of plasma drug concentration and time 0 to infinity and is estimated as the area under the plot of plasma concentration against time 0 to infinity after drug administration. Blood samples collected at designated time points will be used to determine the AUC0-inf of ISL.
AUC0-last of ISL | At designated time points up to ~30 days
  AUC0-last is defined as the area under the concentration-time curve from time zero to time of last measurable concentration of ISL. Blood will be collected at designated time points to determine the AUC0-last of ISL.
Cmax of ISL | At designated time points up to ~30 days
  Cmax is the maximum concentration of the drug observed in plasma. Blood samples collected at designated time points will be used to determine Cmax of ISL.

SECONDARY OUTCOMES:
Number of participants who experienced an adverse event (AE) | Up to ~44 days
  An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. The number of participants with an adverse event will be reported.
Number of participants who discontinued study intervention due to an AE | Up to ~30 days
  An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. The number of participants who discontinue study intervention due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion (Site 0001), Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com